CLINICAL TRIAL: NCT03756194
Title: 'Culture-Aware Robots and Environmental Sensor Systems for Elderly Support' (CARESSES) - Testing and Evaluation Phases
Brief Title: CARESSES Testing and Evaluation Phases
Acronym: CARESSES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Bedfordshire (Other)
Collaborators: Università degli Studi of Genova (Unknown); Örebro University, Sweden (Other); Middlesex University (Other); SoftBank Robotics Europe (Unknown); Advinia Health Care limited (Unknown); Japan Advanced Institute of Science and Technology (Unknown); Nagoya University (Other); Chubu University (Unknown)
Responsible Party: Principal Investigator, Dr Chris Papadopoulos, Principal lecturer in Public Health, University of Bedfordshire
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CARESSES No 737858
Record Dates: First submitted 2018-11-19; First posted 2018-11-28 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Aging
Keywords: Aged; Elders; Robotics; Cultural competence; Quality of life; Loneliness; Technology acceptance; Social robotics; Informal caregiver; Homes for the aged

STUDY DESIGN:
Who Masked: Participant
Masking Description: The researchers and technical staff supporting the experiments are unable to be blinded. Therefore, a single blind masking strategy will be used meaning that the participants and their carers (apart from the control arm 2) will be left unaware of what group they have been allocated to and what type of the CARESSES robot they will be interacting with.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental (Experimental): Participants will utilize the socially-assistive robot with a CARESSES cultural competence solution during 6 sessions (3 times per week, e.g., Monday, Wednesday, and Friday; for a total of 2 weeks) of 3 hours at a time.
  Baseline and follow-up assessments will be conducted prior to the beginning of the trials and shortly after the end of the last session accordingly.
  Interventions: Device: Socially-assistive Pepper robot with a CARESSES cultural competence solution
- Control arm 1 (Other): Participants will utilize the socially-assistive control robot with an alternative CARESSES solution during 6 sessions (3 times per week, e.g., Monday, Wednesday, and Friday; for a total of 2 weeks) of 3 hours at a time.
  Baseline and follow-up assessments will be conducted prior to the beginning of the trials and shortly after the end of the last session accordingly.
  Interventions: Device: Socially-assistive control Pepper robot with an alternative CARESSES solution
- Control arm 2 (No Intervention): Participants will be receiving conventional human care with no robot intervention.
  Baseline assessments will be conducted as soon as participants are recruited and allocated to the study arm. Follow-up assessments will be conducted in two weeks after the baseline data collection.

INTERVENTIONS:
Device: Socially-assistive Pepper robot with a CARESSES cultural competence solution — Week 1. On the first day, training will be provided to the participants enabling them to familiarise themselves with the robot's functionalities. The robot will be culturally aware i.e., it will be aware of the participants' cultural background prior to the testing commencing. As such, it will pre-load the appropriate CKB and apply this during its time with the participants. During the next two sessions, the robot will interact and provide culturally-competent assistance, however, it will not learn and adjust to the participants' individual cultural values and preferences.
  Week 2. The participants will again utilize the robot for three days, but it now will learn from the responses it receives from them, consequently interacting in a culture-specific personalised way.
  Arms: Experimental
Device: Socially-assistive control Pepper robot with an alternative CARESSES solution — Week 1. On the first day, training will be provided to the participants enabling them to familiarise themselves with the robot's functionalities. During the next two sessions, the CARESSES control robot will not be culturally aware: it will pre-load a generic and more limited CKB that is not tailored for anyone's cultural profile. It will also not learn and adjust to the participants' values and preferences.
  Week 2. Participants will again utilize the robot for three days, but the CARESSES control robot will now be configured to be able to learn and adapt to the individual's particular profile. This robot's learning will not include propagation: improving its cultural knowledge base in one area will not also automatically lead to knowledge improvements in other related areas. This robot will possess the same full suite of functions as the CARESSES robot although will be less likely to offer these in a culturally appropriate way.
  Arms: Control arm 1

SUMMARY:
The aim of this study is to conduct and evaluate a controlled experimental trial aimed at exploring whether, to what extent and how a socially-assistive Pepper robot that operates on a unique CARESSES cultural competence solution can produce better health and well-being related outcomes among older adults residing in long stay care homes (and their informal carers) compared to a control socially-assistive Pepper robot with an alternative CARESSES solution, as well as care as usual.

DETAILED DESCRIPTION:
The objective of the "Culture-Aware Robots and Environmental Sensor Systems for Elderly Support' (CARESSES) project is to build culturally competent robots that are able to re-configure their way of acting and speaking when offering a service to a person they are assisting, and match his / her culture, customs and etiquette. This study will test and evaluate robots that have been configured to provide a culturally-competent care to older adults residing in care homes. It is hypothesised that by introducing robots, which are more sensitive to the user's needs and able to adapt to his / her cultural background, the CARESSES' innovative solution will offer a safe, reliable and intuitive system that fosters independence and autonomy, improves quality of life of older adults, and also reduces informal carer's burden. The methodology adopted to develop this culturally competent solution is based on the principles of Transcultural Nursing, specifically on Hofstede's Cultural dimensions theory (for describing general cultural characteristics at national level) and on Papadopoulos, Tilki and Taylor's model of cultural competence.

At the heart of the CARESSES software is a cultural knowledge base (CKB) that stores all the required information about the user and his / her cultural background. CKB was developed using the guidelines provided by the experts in Transcultural Nursing, who identified through field observations differences and similarities between individuals within three cultural groups (i.e. White-English, Indian and Japanese) in order to avoid as much as possible stereotyping and to provide suggestions regarding how likely culturally-specific behaviours are valid for an individual belonging to the cultural group.

The study will employ a mixed method (qualitative and quantitative) single-blind, controlled before-and-after experimental design with two testing sites (UK and Japan), in which participants will either be purposefully allocated to an experimental arm (who will receive and be assisted by the CARESSES robot), control arm 1 (who will receive and be assisted by the control CARESSES robot) or control arm 2 (who will receive care as usual). Between and within subjects comparisons will be used to evaluate whether and how the assistance of a CARESSES Pepper robot improves health and well-being related outcomes among care home residents and their informal carers. Eligible older adults from three cultural groups (White-English, Indian and Japanese) will be recruited from the UK-based (White-English and Indian cultural backgrounds only) and Japanese-based testing sites. Additionally, the participants will be requested to nominate up to three informal carers of their choice who will also be invited to take part in the study, but to a different degree. After the recruitment, the participants from both sites will then be purposefully allocated to either an experimental arm (UK site: n=10; Japan site: n=5) that will adopt the CARESSES robot, or to a control arm 1 (UK site: n=10; Japan site: n=5) that will adopt the CARESSES control robot, or to control arm 2 (UK site: n=10; Japan site n=5).

In the UK site, each of the arms will include five participants who primarily identify themselves with the White-English culture, and five participants who primarily identify themselves with the Indian culture. In the Japan site, three arms will only include participants who primarily identify themselves with the Japanese culture. The participants allocated to the control arm 2 will engage in testing first, followed by the control arm 1 and then the experimental arm. Testing will occur on two participants at any one time in the UK site, and on one participant in the Japan site. Each participant will adopt a Pepper robot over a period of two weeks.

Prior to commencing the full-scale study, a pre-trial feasibility pilot will be conducted aimed at assessing the feasibility and acceptability of the screening, recruitment and evaluation procedures, as well as identifying and tackling any technical issues associated with the implementation of the CARESSES robot within a care home. One resident, who primarily identifies himself / herself with the White-English culture and one informal carer will be invited to take part in the pilot study. The evaluation procedure will take place in a condensed format across one week (9 hours) rather than two weeks (18 hours) as during the full-scale study.

ELIGIBILITY:
Inclusion Criteria (Older Adults):

* Aged ≥ 65 years.
* Reside in an eligible Advinia care home in the UK or within the HISUISUI facility in Japan.
* Reside in a single occupancy bedroom / bedroom area.
* Identify themselves as primarily belonging to the White-English or Indian cultures (UK site only), or Japanese culture (Japan site only).
* Unlikely to express aggression towards themselves, the robot, and/or the researcher (as assessed by the interRAI- Long Term Care Facility (LTCF) tool Aggressive Behaviour Scale (ABS) < 1).
* Have the cognitive ability to participate in the study (as assessed by the interRAI-LTCF tool Cognitive Performance Scale (CPS) ≤ 2).
* Unlikely to fall ill and be hospitalized during study period (as assessed by the FRAIL-NH scale ≤ 10)
* Verbally able to communicate in and understand English (UK site only) or Japanese (Japan site only).

Exclusion Criteria:

* Aged < 65 years.
* Reside in multiple-occupancy bedrooms (UK site only)
* Do not identify themselves as primarily belonging to the Indian, White-English or Japanese culture.
* Likely to express aggression towards themselves the robot, and/or the researcher (as assessed by the interRAI-LTCF tool ABS ≥ 1).
* Do not have sufficient cognitive ability to participate in the study (as assessed by the interRAI-LTCF tool CPS > 2).
* Likely to fall ill and be hospitalized during study period (as assessed by the FRAIL-NH scale > 10)
* Not able to communicate in and understand English (UK site only) or Japanese (Japan site only).

Inclusion criteria (Informal carers)

* Aged ≥18 years.
* Have visited the participant in the care home within the past 3 months.
* Provide any type of informal help, care and/or support to the participant.
* Are a relative, partner, friend or neighbour who has a significant personal relationship with the participant.
* Are not paid or officially employed to provide care to the participant.
* Able to communicate in and understand English (UK site) or Japanese (Japanese site).

Exclusion criteria (Informal carers)

* Aged < 18 years.
* Have not visited the participant in the care home within the past 3 months.
* Not able to verbally communicate in and understand English (UK site only) or Japanese (Japan site only).
* Are formally paid to provide care to the participant.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-02-15 (Actual); Primary Completion 2019-10-31 (Estimated); Study Completion 2020-01-31 (Estimated)

PRIMARY OUTCOMES:
Cultural Competence Assessment Tool -Robotics (CCATool-Robotics): change in perceptions of the robot's cultural competency when assistance provided with and without personalisation. | Two sessions, approximately 15 minutes each in length
  The measurement tool is an adaptation of the RCTSH Cultural Competence Assessment Tool (CCATool; Papadopoulos, Tilki, and Lees, 2004). The current tool is designed to measure older adults' perceptions of the CARESSES robot's cultural awareness, cultural knowledge, cultural sensitivity, and cultural competence. The tool comprises of 28 statements that participants use to rate their level of agreement with.

SECONDARY OUTCOMES:
Short Form (36) Health Survey (SF-36 | Two sessions, approximately 20 minutes each in length
  The SF-36v2 (Hays, Sherbourne, & Mazel, 1993) is a multi-purpose, short-form health survey with 36 questions proven to be useful in surveys of general and specific populations, including older adults. It measures the following eight dimensions: general health, bodily pain, emotional role limitation, physical role limitation, mental health, vitality, physical functioning and social functioning. Each dimension score has values between 0 and 100, in which 0 means dead and 100 perfect health.
The Zarit Burden Inventory (ZBI) | Two sessions, approximately 5 minutes each in length
  A 22-item self-report inventory is aimed at evaluating subjective care burden among informal carers (Zarit, Reever, & Bach-Peterson, 1980). Its validity and reliability have been widely established. The scale items examine burden associated with functional / behavioural impairments and care situations. Each item is scored on a 5-point Likert Scale ranging from "never" to "nearly always present." A total score is obtained with higher scores indicting higher care burden among informal carers.
Short form University of California Los Angeles (UCLA) Loneliness Scale (ULS-8) | Two sessions, approximately 8 minutes each in length
  Loneliness will be measured using the Short-Form Measure of Loneliness (Hays & DiMatteo, 1987). The scale is comprised of eight items to assess loneliness ("I lack companionship", "There is no one I can turn to", "I am an outgoing person", "I feel left out", "I feel isolation from others", "I can find companionship when I want it", "I am unhappy being so withdrawn", "People are around me but not with me") using a 4-point Likert scale with values ranging from "never" to "always". To obtain a total score, all values are added up, and the higher scores are, the bigger feeling of loneliness may be presumed.
Questionnaire for user interface satisfaction (QUIS) | One session, approximately 10 minutes in length
  A measure of overall system satisfaction along six scales, and hierarchically organized measures of eleven specific interface factors (screen factors, terminology and system feedback, learning factors, system capabilities, technical manuals, on-line tutorials, multimedia, voice recognition, virtual environments, internet access, and software installation; Chin, Diehl, & Norman, 1988). Each area measures the users' overall satisfaction with that facet of the interface, as well as the factors that make up that facet, on a 9-point scale. The questionnaire is designed to be configured according to the needs of each interface analysis by including only the sections that are of interest to the user. Taking into consideration the context of the current study, "the software" is replaced by "the robot" where required.
Negative attitudes towards robots scale (NARS) | Two sessions, approximately 5 minutes each in length
  This scale assesses participants' attitudes towards robots (Nomura, Kanda, Suzuki, & Kato, 2004). NARS is comprised of 14 items scored on a 5-point Likert Scale (1= I completely disagree; 5=I completely agree), which in turn belong to three subscales: S1 measures "situations of interaction with robots," S2 measures "social inﬂuence of robots," and S3 measures "emotions in interaction with robots".
Older adults' perceptions of the robot's cultural competence and overall experience | One session, approximately 5 minutes each in length
  Semi-structured interviews with older adults from the experimental group will be conducted to elicit their perceptions of the robot's cultural competence; acceptability of and satisfaction with the robot interactions; quality of service provided; and impact the robot had upon their health and well-being, independence and autonomy.
Informal carers' experience of using the robot | One session, approximately 20 minutes each in length
  Semi-structured interviews with informal carers' from the experimental group will be conducted to receive their feedback on whether and how the robot reduced any feelings of carer burden and stress; their perceptions of whether and how the robot impacted upon the quality of life of both themselves and the resident; and perceptions regarding the robot's ease of use when interacting with it.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Sgorbissa, ASSOC PROFESSOR, Principal Investigator — Università di Genova
Locations (1):
- University of Bedfordshire, Luton, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Papadopoulos C, Hill T, Battistuzzi L, Castro N, Nigath A, Randhawa G, Merton L, Kanoria S, Kamide H, Chong NY, Hewson D, Davidson R, Sgorbissa A. The CARESSES study protocol: testing and evaluating culturally competent socially assistive robots among older adults residing in long term care homes through a controlled experimental trial. Arch Public Health. 2020 Mar 20;78:26. doi: 10.1186/s13690-020-00409-y. eCollection 2020. PMID 32206312
- See also: Related Info — http://caressesrobot.org/en/